CLINICAL TRIAL: NCT05888818
Title: The Effect of Cold Application on Nausea and Vomiting in the Early Postoperative Period - Randomized Controlled Study
Brief Title: The Effect of Cold Application on Nausea and Vomiting in the Early Postoperative Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Nigar Ak Turkis, Doctoral Candidate in Surgical Nursing Science, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/16-08
Record Dates: First submitted 2023-05-03; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Local Application/Packing Too Cold; Patient Satisfaction; Postoperative Nausea and Vomiting
Keywords: Nausea and vomiting after surgery,cold application methods,nursing care after surgery,alternative and complementary methods,postoperative care,cholecystectomy; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction; Postoperative Nausea and Vomiting; Nausea

STUDY DESIGN:
Intervention Model Description: There is an experimental and a control group.The distribution of the patients to the groups was made according to the random numbers table obtained by using the index formulas and randomly in the excel program in the web environment.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold application group (Experimental): A cold application (with a cold gel pack) will be applied to the upper part of the neck for 5 minutes.
  Interventions: Other: Cold application
- standard treatment (No Intervention): No application will be made and the presence of nausea, severity, vomiting and vital signs will be measured after 5 minutes.

INTERVENTIONS:
Other: Cold application — A cold application (with a cold gel pack) will be applied to the upper part of the neck for 5 minutes.
  Arms: cold application group

SUMMARY:
As a result of the literature review, it has been seen that it has not yet been clarified whether cold application methods are effective on postoperative nausea and vomiting, and academic studies on this subject are needed.

The aim of the planned study was to conduct a randomized controlled experimental study to evaluate the effect of the cold application method on nausea and vomiting and the need for antiemetic drugs in the early postoperative period.

The research hypotheses are as follows:

H1:Cold application method reduces nausea and vomiting in the early postoperative period.

H1:The cold application method reduces the need for antiemetic drugs in the early postoperative period.

H1:Cold application method in the early postoperative period increases patient satisfaction.

Condition or disease:

Postoperative nausea and vomiting,Postoperative antiemetic use status,Patient satisfaction,Effects of cold application method

Intervention/treatment:

There is an intervention group in which the cold application method is applied.

DETAILED DESCRIPTION:
The aim of the planned study was to conduct a randomized controlled experimental study to evaluate the effect of the cold application method on nausea and vomiting and the need for antiemetic drugs in the early postoperative period.

The population of the study will consist of patients who are planned to undergo laparoscopic cholecystectomy under general anesthesia in the Department of General Surgery, Zonguldak Bülent Ecevit University Health Practice and Research Center between October 2022 and October 2024.Çalışmanın örneklemini laparoskopik kolesistektomi planlanan, dahil edilme kriterlerini karşılayan ve çalışmaya katılmaya gönüllü olan hastalar oluşturacaktır.

As a result of the GPower power analysis, it was calculated that at least 60 people (at least 30 people for each group) who met the inclusion criteria of the research should be taken in order to obtain 80% power at the 95% confidence interval for the d=0.8 effect size.

Data collecting:

The collection of research data will be carried out in three stages.

1. stage:Patients scheduled for laparoscopic cholecystectomy who have undergone hospitalization will be evaluated in terms of their eligibility for inclusion criteria, and eligible patients will be invited to participate in the study.The purpose of the research will be explained to the patients, the informed consent form will be read, written and verbal consent will be obtained and a copy of the form will be given to the patients.Then, the patient information data collection form and Apfel risk score will be filled with face-to-face interview technique, and the answers given by the patients will be recorded.
2. stage: The surgery will be held in the recovery room.While the patients in the intervention group are in the recovery room after the surgery, their routine applications will be made and the state of consciousness and alertness will be checked.After the application, the presence of nausea, severity, vomiting status, vital signs (blood pressure, pulse, respiratory rate, body temperature) will be measured.Then, a cold application (with a cold gel pack) will be applied to the nape area for 5 minutes.Presence of nausea, severity, vomiting status, vital signs will be re-measured immediately after the application.Antiemetic drug use and opioid drug use will be questioned.
3. stage:Presence, severity and presence of nausea will be re-evaluated at the 2nd and 6th hours of the experimental and control group patients.Antiemetic drug use and opioid drug use will be questioned.Patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Those who will undergo elective surgery
* Attempting laparoscopic cholecystectomy
* Those between the ages of 18-65
* Those who will receive general anesthesia
* Not allergic to cold
* Body temperature ≥36°C
* ASA I and ASA II class
* Those with an Apfel risk score of 2 and above
* Postoperative nausea severity of 2 and above
* Without chronic disease
* Neurological problems
* No problem communicating,• No hearing and vision problems
* Being conscious, awake and oriented after surgery,
* Patients who volunteer to participate in the study will be included in the study

Exclusion Criteria:

* Those who are allergic to cold
* Body temperature <36°C,
* Those who have a disability, incision and surgical procedure around the head and neck
* Having chronic illness
* Having neurological problems
* Having nasogastric tube
* Postoperatively conscious, awake and not oriented,
* Not eligible for inclusion criteria and
* Patients who do not volunteer to participate in the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Determining the mean scores of the experimental and control groups from the nausea numerical scale | two year
  Nausea Numerical Scale There are numbers from 0 to 10 on the scale.The scale is explained to the patients and asked to choose the number between 0 and 10 that best reflects their nausea.
  Zero usually indicates 'no nausea' while 10 represents 'unbearable nausea'. Evaluation will be made in the recovery room after the surgery, then at the 2nd and 6th hours.
Determination of patient satisfaction of the experimental and control groups | two year
  The patient satisfaction scale is used to evaluate patient satisfaction.It consists of numbers between "0" and "10" to determine the satisfaction level of the patients after the A value of zero indicates "no satisfaction" with the practice, while a value of ten indicates "a lot of satisfaction". Satisfaction scale will be evaluated at the 6th hour after the surgery.
Antiemetic use status of the groups | two year
  The patients' use of antiemetics after surgery will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Nigar AK TURKİS, PhD student, Principal Investigator — Zonguldak Bulent Ecevit University,PhD student
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No